CLINICAL TRIAL: NCT00005619
Title: Detection of Hairy Cell Leukemia Minimal Residual Disease: Detection by Flow Cytometry
Brief Title: Analysis of Blood and Bone Marrow to Detect Residual Disease in Patients With Previously Treated Hairy Cell Leukemia
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: LoAnn Peterson, MD, Northwestern University
Other Study IDs: NU 97Z3; NU-97Z3; NCI-G00-1754
Record Dates: First submitted 2000-05-02; First posted 2004-07-19 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Leukemia
Keywords: progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Hairy Cell | interventions — Polymerase Chain Reaction; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Genetic: polymerase chain reaction
Other: flow cytometry
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Diagnostic procedures that detect residual disease may predict disease relapse in patients who have hairy cell leukemia.

PURPOSE: Diagnostic trial to determine the effectiveness of analyzing blood and bone marrow to detect residual disease in patients who have previously treated hairy cell leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the sensitivity of flow cytometry, immunohistochemistry, and polymerase chain reaction in detecting minimal residual disease following therapy with cladribine in patients with hairy cell leukemia.

OUTLINE: Blood and bone marrow samples are obtained from patients at time of bone marrow biopsies to assess minimal residual disease using flow cytometry, immunohistochemistry, and polymerase chain reaction. Patients are followed for 2 years or until disease relapse.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study over 12-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Clinically documented hairy cell leukemia Active or in remission Must have received prior cladribine and be undergoing bone marrow biopsies as follow up

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior chemotherapy following prior cladribine Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a documented diagnosis of hairy cell leukemia who are undergoing routine bone marrow boipsy/aspiration and peripheral blood collection.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2000-02; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loann C. Peterson, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States